CLINICAL TRIAL: NCT05596578
Title: Role of Intrapulmonary Lymph Nodes in Patients With NSCLC and Visceral Pleural Invasion
Status: Recruiting | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Fabrizio Minervini, Staff Surgeon Thoracic Surgery, Luzerner Kantonsspital
Other Study IDs: 2022.10.Thx
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer; Lymph Node Metastasis
MeSH Terms: conditions — Lung Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Patients who underwent an anatomical resection for NSCLC <3 cm (lobectomy, bilobectomy, segmentectomy) with samples from the intrapulmonary stations 12, 13, and 14 lymph nodes and resection of lymph nodes station 10 and 11 during hilar separation.

SUMMARY:
Background: Lung cancer is the leading cause of cancer related death worldwide. More than 80% of all lung tumors are Non-Small Cell Lung Cancers (NSCLC). Lymph node staging has a prognostic value and is crucial to establish the optimal treatment strategy in individual patients. It remains unknown whether dissecting the intrapulmonary lymph nodes (stations 13 and 14) is necessary for accurate staging and prognostication. Although suggested by several guidelines, these peripheral lymph nodes are not routinely examined in clinical routine for several reasons. Moreover, the prognostic significance of the visceral pleural invasion is controversial. Some studies showed a negative impact on OS and DFS in patients with histologic proved visceral pleura invasion.

The mechanism to explain this negative effect is not fully understood. Given that the visceral pleura is very rich in lymphatic vessels, with an intercommunicating "network" arranged over the lung surface and penetrating into the lung parenchyma to join the bronchial lymph vessels with drainage to the various hilar nodes, we assume that the worse OS and DFS observed in these patients could be explained with the presence of metastatic lymph nodes (Station 13-14) that are not routinely examined. Methods: This is a prospective, multicenter study based on ad-hoc created prospectively database. The incidence of N1 lymph node metastasis overall and the incidence of metastasis to the different lymph node stations (Hilar 10/11, Lobar 12, Sublobar 13/14) will be calculated by dividing the number of the respective events by the patient years separately. To investigate the association between visceral pleural invasion and the presence of metastatic lymph nodes univariate and multivariate logistic regression models will be fitted to the data.

Discussion: The primary outcome is to investigate the incidence of N1 metastases (especially stations 12,13,14) and his relationship with visceral pleural invasion. The secondary outcomes is to evaluate the impact of N1 metastases and/or visceral pleural invasion on long-term outcomes (OS and DFS) along with incidence and pattern of recurrence. DFS is defined as the time of surgical intervention to tumor recurrence or death, and OS is defined as the time of surgical intervention to death

ELIGIBILITY:
Inclusion Criteria:

* Anatomical resection for NSCLC <3 cm (lobectomy, bilobectomy, segmentectomy)
* Samples from the intrapulmonary stations 12, 13, and 14 lymph nodes
* Resection of lymphnodes station 10 and 11 during hilar separation.
* R0 resection

Exclusion Criteria:

* Prior or synchronous lung cancer
* pN2
* Pneumonectomy
* R1/R2 resection
* M1
* Neoadjuvant treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients recorded prospectively in the database from January 2023 to December 2024 that meet the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 958 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
N1 | January 2023-December 2024
  Overall incidence of N1 pathological lymph nodes (Hilar 10/11, Lobar 12, Sublobar 13/14)
VPI | January 2023-December 2024
  Incidence of N1 pathological lymph nodes (Hilar 10/11, Lobar 12, Sublobar 13/14) in patients with pathological evidence of visceral pleural invasion

SECONDARY OUTCOMES:
OS | January 2023- December 2029
  Overall Survival (1-3-5 Years)
DFS | January 2023-December 2029
  Disease free survival (1-3-5 Years)
Tumor recurrence | January 2023-December 2029
  pattern : local, regional, distant

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Luzern, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang H, Wang T, Hu B, Pan C. Visceral pleural invasion remains a size-independent prognostic factor in stage I non-small cell lung cancer. Ann Thorac Surg. 2015 Apr;99(4):1130-9. doi: 10.1016/j.athoracsur.2014.11.052. Epub 2015 Feb 20. PMID 25704861
- [Background] Bi L, Zhang H, Ge M, Lv Z, Deng Y, Rong T, Liu C. Intrapulmonary lymph node (stations 13 and 14) metastasis in peripheral non-small cell lung cancer. Medicine (Baltimore). 2021 Jul 9;100(27):e26528. doi: 10.1097/MD.0000000000026528. PMID 34232188
- [Background] Seok Y, Lee E. Visceral Pleural Invasion Is a Significant Prognostic Factor in Patients with Partly Solid Lung Adenocarcinoma Sized 30 mm or Smaller. Thorac Cardiovasc Surg. 2018 Mar;66(2):150-155. doi: 10.1055/s-0036-1586757. Epub 2016 Aug 12. PMID 27517168
- [Background] Park S, Cho S, Yum SW, Kim K, Jheon S. Comprehensive analysis of metastatic N1 lymph nodes in completely resected non-small-cell lung cancer. Interact Cardiovasc Thorac Surg. 2015 Nov;21(5):624-9. doi: 10.1093/icvts/ivv209. Epub 2015 Aug 4. PMID 26242319
- [Background] Wightman SC, Lee JY, Ding L, Atay SM, Shemanski KA, McFadden PM, David EA, Kim AW. Adjuvant chemotherapy for visceral pleural invasion in 3-4-cm non-small-cell lung cancer improves survival. Eur J Cardiothorac Surg. 2022 Jun 15;62(1):ezab498. doi: 10.1093/ejcts/ezab498. PMID 35325098
- [Background] Fibla JJ, Cassivi SD, Brunelli A, Decker PA, Allen MS, Darling GE, Landreneau RJ, Putnam JB. Re-evaluation of the prognostic value of visceral pleura invasion in Stage IB non-small cell lung cancer using the prospective multicenter ACOSOG Z0030 trial data set. Lung Cancer. 2012 Dec;78(3):259-62. doi: 10.1016/j.lungcan.2012.09.010. Epub 2012 Oct 3. PMID 23040416
- [Background] Nitadori JI, Colovos C, Kadota K, Sima CS, Sarkaria IS, Rizk NP, Rusch VW, Travis WD, Adusumilli PS. Visceral pleural invasion does not affect recurrence or overall survival among patients with lung adenocarcinoma </= 2 cm: a proposal to reclassify T1 lung adenocarcinoma. Chest. 2013 Nov;144(5):1622-1631. doi: 10.1378/chest.13-0394. PMID 23807749
- [Derived] Minervini F, Kestenholz P, Bertoglio P, Li A, Nilius H. Role of intrapulmonary lymph nodes in patients with NSCLC and visceral pleural invasion. The VPI 1314 multicenter registry study protocol. PLoS One. 2023 May 4;18(5):e0285184. doi: 10.1371/journal.pone.0285184. eCollection 2023. PMID 37141291